CLINICAL TRIAL: NCT05810233
Title: The Effect of Vitamin C on the Skin Prick Test Wheal Reaction
Brief Title: Effect of Vitamin C on Allergy Skin Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, ANEEZA KHAIRIYAH WAN HAMIZAN, Associate Professor, Dr, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: JEP-2023
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Rhinitis, Allergic; Allergy
Keywords: ascorbic acid; skin prick test; vitamin C; antihistamine
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Participant assigned to only one intervention per arm either vitamin C or placebo tablets
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Tablets will be despensed by a research assistant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Commercially available Tablet Vitamin C 1000mg per day for 7 days
  Interventions: Dietary Supplement: Ascorbic acid 1000mg
- Placebo (Placebo Comparator): Glucose chewable table 1x per day for seven days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ascorbic acid 1000mg — Health supplement
  Other Names: VItamin C
  Arms: Vitamin C
Other: Placebo — Glucose chewable tablet without any ascorbic acid
  Arms: Placebo

SUMMARY:
This study will assess the effect of taking vitamin C on allergy skin test.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is an Immunoglobulin E (IgE) mediated inflammation of the nasal cavity. House dust mite is the most common causative allergen. The skin prick test is the preferred method to confirm allergy. This test is interpreted by measuring the skin wheal reaction in response to allergen application and histamine. Prior studies have shown that Vitamin C may have antihistamine effect that may reduce the wheal reaction in skin prick test thus cause difficulties to interpret the results. Current guidelines do not recommend cessation of vitamin C prior to skin prick test. This will require further study in order to further understand the effect of vitamin C in commercially available dose on the skin prick test wheal reaction. In this randomized placebo controlled trial, consecutive participant visiting the ENT clinic with allergic rhinitis and prior positive skin prick test towards dust mite will be screened for inclusion and exclusion criteria. Participants will either receive vitamin C 1000mg daily for 7 days or placebo. The skin prick test will be performed after one week of intervention and the area of the wheal reaction area (mm2) and longest diameter (mm) recorded. This will be compared between the two groups. The expected outcome is that participants with oral supplementation of vitamin C will have reduced SPT wheal reaction compared to placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Participants above 18-years old
* Participants with history at least 2 symptoms of rhinitis triggered by dust
* Positive SPT to Dermatophagoides pteronyssinus with wheal reaction of at least 5 mm done within the past 1 year.

Exclusion Criteria:

* Prior skin prick test result form do not include a tracing of the wheal reaction.
* Prior skin prick test was not performed in HCTM.
* Participants who are actively smoking or who have smoked cigarette or vaped in the past 6 months
* Participants with skin conditions affecting the volar aspects of the arm.
* Participants on beta-blockers
* Participants contraindicated for skin prick test (pregnancy, history of anaphylaxis, poorly controlled asthma)
* Participants on long term supplements (multivitamin, traditional supplement)
* Participants contraindicated for vitamin c (vitamin c allergy, kidney dysfunction, history of kidney or bladder stones, hyperuricemia, thalassemia, G6PD deficiency, sickle cell disease, hamatochromatosis)
* Participants at risk of vitamin C deficiency (hyperthyroidism, elderly, beastfeeding, diarrhoea, restricted diet secondary to inflammatory bowel disease, anorexia or cancer)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Skin prick test wheal area of vitamin C group compared to placebo | Day 8
  Skin wheal reaction is measured using computer software. Day 8 wheal area of vitamin C group compared to placebo.

SECONDARY OUTCOMES:
Skin prick test wheal reaction at day 8 of intevention compraed to prior skin prick test done as standard of care | Day 8
  Skin wheal reaction are is measured from prior skin test record (baseline) and at day 8 skin test repeated and measured. Area at day 7 - baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Aneeza K W Hamizan, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Mukhriz, Cheras, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared if journal is required

REFERENCES:
- [Background] Skoner DP. Allergic rhinitis: definition, epidemiology, pathophysiology, detection, and diagnosis. J Allergy Clin Immunol. 2001 Jul;108(1 Suppl):S2-8. doi: 10.1067/mai.2001.115569. PMID 11449200
- [Background] Fortner BR Jr, Danziger RE, Rabinowitz PS, Nelson HS. The effect of ascorbic acid on cutaneous and nasal response to histamine and allergen. J Allergy Clin Immunol. 1982 Jun;69(6):484-8. doi: 10.1016/0091-6749(82)90171-3. PMID 7076989